CLINICAL TRIAL: NCT03068455
Title: A Phase 3, Randomized Study of Adjuvant Immunotherapy With Nivolumab Combined With Ipilimumab Versus Nivolumab Monotherapy After Complete Resection of Stage IIIb/c/d or Stage IV Melanoma
Brief Title: An Investigational Immuno-therapy Study of Nivolumab Combined With Ipilimumab Compared to Nivolumab by Itself After Complete Surgical Removal of Stage IIIb/c/d or Stage IV Melanoma
Acronym: CheckMate 915
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CA209-915; 2016-003729-41 (EudraCT Number)
Record Dates: First submitted 2017-02-27; First posted 2017-03-01 (Actual); Results first posted 2021-07-22 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-08

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- nivolumab + ipilimumab (Experimental): Specified Dose on Specified Days
  Interventions: Biological: nivolumab; Biological: ipilimumab
- nivolumab (Experimental): Specified Dose on Specified Days
  Interventions: Biological: nivolumab

INTERVENTIONS:
Biological: nivolumab — Specified Dose on Specified Days
  Other Names: Opdivo; BMS-936558
Biological: ipilimumab — Specified Dose on Specified Days
  Other Names: Yervoy; BMS-734016
  Arms: nivolumab + ipilimumab

SUMMARY:
The purpose of this study is to determine whether an investigational immunotherapy Nivolumab, when combined with Ipilimumab, is more effective than Nivolumab by itself, in delaying the return of cancer in patients who have had a complete surgical removal of stage IIIb/c/d or stage IV Melanoma

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Completely surgically resected stage IIIb/c/d or stage IV melanoma within 12 weeks of participation in study.
* Must have full activity or, if limited, must be able to walk and carry out activities such as light house work or office work
* No prior anti-cancer treatment for melanoma (except surgery for the melanoma lesion(s) and/or except for adjuvant radiation therapy (RT) after neurosurgical resection for central nervous system (CNS) lesions)

Exclusion Criteria:

* History of uveal melanoma
* Patients with active, known or suspected autoimmune disease
* Prior treatment with interferon (if complete < 6 months prior to participation in study), anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1844 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2021-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (120):
- United States (33):
  - University of Arizona Cancer Center, Tucson, Arizona
  - The Angeles Clinic & Research Institute, Los Angeles, California
  - California Pacific Medical Center, San Francisco, California
  - University Of Colorado, Aurora, Colorado
  - Georgetown University Med Ctr, Washington D.C., District of Columbia
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - UF Health Cancer Center at Orlando Health, Orlando, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute, Atlanta, Georgia
  - University Of Chicago, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Oncology Specialists, S.C., Park Ridge, Illinois
  - Mass General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University Of Michigan Health System, Ann Arbor, Michigan
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University School Of Medicine, St Louis, Missouri
  - NYU Langone Medical Center, New York, New York
  - Memorial Sloan Kettering Nassau, New York, New York
  - Carolinas Med Ctr, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Providence Cancer Center Oncology And Hematology Care, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - St. Luke's University Health Network, Easton, Pennsylvania
  - Local Institution, Nashville, Tennessee
  - Texas Oncology Sammons Cancer Center, Dallas, Texas
  - Md Anderson Can Cnt, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - University Of Virginia Health System, Charlottesville, Virginia
  - Inova Melanoma and Skin Cancer Center, Fairfax, Virginia
  - University Of Washington Cancer Care Alliance, Seattle, Washington
- Australia (11):
  - Local Institution, North Sydney, New South Wales
  - Local Institution, Waratah, New South Wales
  - Local Institution, Westmead, New South Wales
  - Local Institution, Greenslopes, Queensland
  - Local Institution, Southport, Queensland
  - Local Institution, Woolloongabba, Queensland
  - Local Institution, Adelaide, South Australia
  - Local Institution, Box Hill, Victoria
  - Local Institution, Melbourne, Victoria
  - Local Institution, Nedlands, Western Australia
  - Local Institution, Subiaco, Western Australia
- Austria (2):
  - Local Institution, Graz
  - Local Institution, Vienna
- Belgium (3):
  - Local Institution, Brussels
  - Local Institution, Ghent
  - Local Institution, Liège
- Brazil (9):
  - Local Institution, Salvador, Estado de Bahia
  - Local Institution, Belo Horizonte, Minas Gerais
  - Local Institution, Ijuí, Rio Grande do Sul
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Florianópolis, Santa Catarina
  - Local Institution, Barretos, São Paulo
  - Local Institution, São José do Rio Preto, São Paulo
  - Local Institution, Rio de Janeiro
  - Local Institution, São Paulo
- Canada (6):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Local Institution, Montreal, Quebec
  - CHU de Quebec - Universite Laval, Québec, Quebec
- Czechia (4):
  - Klinika komplexni onkologicke pece, Brno
  - Klinika onkologie a radioterapie, Hradec Králové
  - Dermatovenerologicka klinika 3. LF UK a FNKV, Prague
  - Dermatovenerologicka klinika VFN a 1. LF UK, Prague
- France (8):
  - Centre Hospitalier Universitaire Dijon Bocage, Dijon
  - Hopital Claude Huriez, Lille
  - Hopital De La Timone, Marseille
  - Chu Nantes, Nantes
  - Hopital Saint Louis, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif
- Germany (9):
  - Local Institution, Berlin
  - Local Institution, Buxtehude
  - Local Institution, Essen
  - Local Institution, Gera
  - Local Institution, Hanover
  - Local Institution, Heidelberg
  - Local Institution, Lübeck
  - Local Institution, München
  - Local Institution, Tübingen
- Greece (2):
  - Laiko Hospital, Athens
  - Metropolitan Hospital, Athens
- Israel (3):
  - Local Institution, Haifa
  - Local Institution, Jerusalem
  - Local Institution, Tel Litwinsky
- Italy (6):
  - ASST Papa Giovanni XXIII, Bergamo
  - Ospedale Policlinico San Martino, Genova
  - IRCCS Istituto Nazionale Tumori Milano, Milan
  - Istituto Nazionale Tumori Fondazione Pascale, Napoli
  - Istituto Oncologico Veneto IOV, Padua
  - Azienda Ospedaliera Universitaria Senese, Siena
- New Zealand (3):
  - Local Institution, Tauranga, Bay of Plenty
  - Local Institution, Christchurch
  - Local Institution, Dunedin
- Poland (2):
  - Klinika Nowotworow Ukladowych i Uogolnionych, Krakow
  - Klinika Nowotworow Tkanek Miekkich, Kosci i Czerniakow, Warsaw
- Romania (2):
  - Institute Of Oncology "Prof.Dr.Alexandru Trestioreanu" Bucha, Bucharest
  - Sf. Nectarie Oncology Center, Craiova
- Russia (3):
  - Local Institution, Krasnodar
  - Local Institution, Krasnoyarsk
  - Local Institution, Moscow
- Spain (7):
  - Hospital Universitari Germans Trias I Pujol, Badalona-barcelona
  - H. Univ. Vall dHebron, Barcelona
  - Hospital Clinic I Provincial, Barcelona
  - Hospital Gral. Univ. Gregorio Maranon, Madrid
  - Hospital Regional Universitario De Malaga, Málaga
  - Hosp Univ Virgen Macarena, Seville
  - Hospital Universitario Y Politecnico La Fe, Valencia
- Switzerland (2):
  - Local Institution, Lausanne
  - Local Institution, Zurich
- United Kingdom (5):
  - Local Institution, Oxford, Oxfordshire
  - The Beatson West Of Scotland Cancer Centre, Glasgow
  - The Royal Marsden Hospital, London
  - Christie Hospital Nhs Trust, Manchester
  - Royal Marsden Hospital - Surrey, Sutton

REFERENCES:
- [Derived] Long GV, Tang H, Desai K, Wang S, Del Vecchio M, Larkin J, Ritchings C, Huang SP, Baden J, Balli D, Chang H, Fusaro G, Tenney D, Dolfi S, Weber J. Pretreatment and on-treatment ctDNA and tissue biomarkers predict recurrence in patients with stage IIIB-D/IV melanoma treated with adjuvant immunotherapy: CheckMate 915. J Immunother Cancer. 2025 Jul 11;13(7):e012034. doi: 10.1136/jitc-2025-012034. PMID 40645660
- [Derived] Weber JS, Schadendorf D, Del Vecchio M, Larkin J, Atkinson V, Schenker M, Pigozzo J, Gogas H, Dalle S, Meyer N, Ascierto PA, Sandhu S, Eigentler T, Gutzmer R, Hassel JC, Robert C, Carlino MS, Di Giacomo AM, Butler MO, Munoz-Couselo E, Brown MP, Rutkowski P, Haydon A, Grob JJ, Schachter J, Queirolo P, de la Cruz-Merino L, van der Westhuizen A, Menzies AM, Re S, Bas T, de Pril V, Braverman J, Tenney DJ, Tang H, Long GV. Adjuvant Therapy of Nivolumab Combined With Ipilimumab Versus Nivolumab Alone in Patients With Resected Stage IIIB-D or Stage IV Melanoma (CheckMate 915). J Clin Oncol. 2023 Jan 20;41(3):517-527. doi: 10.1200/JCO.22.00533. Epub 2022 Sep 26. PMID 36162037
- [Derived] Yoshino T, Oki E, Misumi T, Kotaka M, Manaka D, Eto T, Hasegawa J, Takagane A, Nakamura M, Kato T, Munemoto Y, Nakamura F, Bando H, Taniguchi H, Sakamoto Y, Shiozawa M, Nishi M, Horiuchi T, Yamagishi H, Sakamoto J, Mizushima T, Ohtsu A, Mori M. Final Analysis of 3 Versus 6 Months of Adjuvant Oxaliplatin and Fluoropyrimidine-Based Therapy in Patients With Stage III Colon Cancer: The Randomized Phase III ACHIEVE Trial. J Clin Oncol. 2022 Oct 10;40(29):3419-3429. doi: 10.1200/JCO.21.02628. Epub 2022 May 5. PMID 35512259
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1844 participants randomized and 1833 treated. Reasons not treated: 1 disease progression; 2 participants withdrew consent; 1 poor/non-compliance; 4 participants no longer met study criteria; 3 not reported
Groups:
- Arm A: Nivo + Ipi: Arm A: nivolumab 240 mg IV Q2 weeks plus ipilimumab 1 mg/kg IV Q6 weeks (for 1 year of study drug treatment)
- Arm B: Nivo: Arm B: nivolumab 480 mg IV Q4 weeks (for 1 year of study drug treatment) with nivolumab placebo on Weeks 3, 7, 11, 15, 19, 23, 27, 31, 35, 39, 43, & 47 and ipilimumab placebo on Weeks 1, 7, 13, 19, 25, 31, 37, 43, & 49
Period: Pre-treatment Period
Arm/Group | Arm A: Nivo + Ipi | Arm B: Nivo
Started (Started = Randomized) | 920 | 924
Completed (Completed = Treated) | 916 | 917
Not Completed | 4 | 7
Not completed — Disease progression | 0 | 1
Not completed — Participant withdrew consent | 1 | 1
Not completed — Poor/non-compliance | 0 | 1
Not completed — Participant no longer meets study criteria | 1 | 3
Not completed — Not reported | 2 | 1
Period: Treatment Period
Arm/Group | Arm A: Nivo + Ipi | Arm B: Nivo
Started (Started = Treated) | 916 | 917
Completed (Completed = Finished treatment period) | 364 | 561
Not Completed | 552 | 356
Not completed — Disease progression | 166 | 208
Not completed — Study drug toxicity | 317 | 104
Not completed — Adverse Event unrelated to study drug | 15 | 7
Not completed — Participant request to stop therapy | 33 | 20
Not completed — Participant withdrew consent | 5 | 10
Not completed — Poor/non-compliance | 3 | 0
Not completed — Participant no longer meets study criteria | 1 | 3
Not completed — Other reasons | 12 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Nivo + Ipi | Arm B: Nivo | Total
Number analyzed (Participants) | 920 | 924 | 1844
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.8 (14.6) | 54.6 (13.7) | 54.2 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 405 | 387 | 792
  Male | 515 | 537 | 1052
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 22 | 44
  Not Hispanic or Latino | 359 | 376 | 735
  Unknown or Not Reported | 539 | 526 | 1065
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 907 | 911 | 1818
  Race: Black or African American | 4 | 1 | 5
  Race: American Indian or Alaska Native | 0 | 1 | 1
  Race: Asian | 3 | 5 | 8
  Race: Other | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Recurrence-free Survival (RFS) - All Randomized Participants
Description: RFS was defined as the time between the date of randomization and the date of first recurrence (local, regional or distant metastasis), new primary melanoma (including melanoma in situ), or death (from any cause), whichever occurred first.
  Median values based on Kaplan-Meier Estimates.
Time Frame: From randomization to Primary Completion Date (up to approximately 3 years)
Population: All randomized participants with completely resected stage IIIb/c/d or stage IV no evidence of disease (NED) melanoma
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Nivo + Ipi | Arm B: Nivo
Number analyzed (Participants) | 918 | 922
Months | NA [NA to NA] — Median not reached as Kaplan-Meier plot did not reach 0.5 probability of recurrence-free survival | NA [NA to NA] — Median not reached as Kaplan-Meier plot did not reach 0.5 probability of recurrence-free survival
Statistical Analysis 1: Comparison: Arm A: Nivo + Ipi vs Arm B: Nivo; Test type: Superiority; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.78 to 1.04] — Stratified Cox proportional hazard model. Hazard Ratio is Nivolumab + Ipilimumab over Nivolumab

2. Primary Outcome: Recurrence-free Survival (RFS) - All Randomized Participants With PD-L1 Expression Level < 1%
Description: RFS was defined as the time between the date of randomization and the date of first recurrence (local, regional or distant metastasis), new primary melanoma (including melanoma in situ), or death (from any cause), whichever occurred first.
  Median based on Kaplan-Meier Estimates.
Time Frame: From randomization to Primary Completion Date (up to approximately 3 years)
Population: All randomized participants with PD-L1 expression level < 1% and with completely resected stage IIIb/c/d or stage IV no evidence of disease (NED) melanoma. PD-L1 expression levels based on Interactive Response Technology (IRT)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Nivo + Ipi | Arm B: Nivo
Number analyzed (Participants) | 347 | 350
Months | 33.15 [22.21 to NA] — Upper limit not calculable as upper CI bound does not cross 50% threshold | 27.63 [19.81 to NA] — Upper limit not calculable as upper CI bound does not cross 50% threshold
Statistical Analysis 1: Comparison: Arm A: Nivo + Ipi vs Arm B: Nivo; Test type: Superiority; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.75 to 1.14] — Stratified Cox proportional hazard model. Hazard Ratio is Nivolumab + Ipilimumab over Nivolumab

3. Secondary Outcome: Overall Survival (OS) - All Randomized Participants
Description: OS is defined as the time between the date of randomization and the date of death. Median based on Kaplan-Meier Estimates.
Time Frame: From randomization to date of death (up to approximately 45 months)
Population: All randomized participants with completely resected stage IIIb/c/d or stage IV no evidence of disease (NED) melanoma
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Nivo + Ipi | Arm B: Nivo
Number analyzed (Participants) | 918 | 922
Months | NA [NA to NA] — Median not reached as Kaplan-Meier plot did not reach 0.5 probability of overall survival | NA [NA to NA] — Median not reached as Kaplan-Meier plot did not reach 0.5 probability of overall survival
Statistical Analysis 1: Comparison: Arm A: Nivo + Ipi vs Arm B: Nivo; Test type: Superiority; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.80 to 1.32] — Stratified Cox proportional hazard model. Hazard Ratio is Nivolumab + Ipilimumab over Nivolumab

4. Secondary Outcome: Overall Survival (OS) - All Randomized Participants With PD-L1 Expression Level < 1%
Description: as for outcome 3
Time Frame: From randomization to date of death (up to approximately 45 months)
Population: All randomized participants with PD-L1 expression level < 1% and with completely resected stage IIIb/c/d or stage IV no evidence of disease (NED) melanoma
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Nivo + Ipi | Arm B: Nivo
Number analyzed (Participants) | 347 | 350
Months | NA [41.72 to NA] — Median not reached as Kaplan-Meier plot did not reach 0.5 probability of overall survival | NA [NA to NA] — Median not reached as Kaplan-Meier plot did not reach 0.5 probability of overall survival
Statistical Analysis 1: Comparison: Arm A: Nivo + Ipi vs Arm B: Nivo; Test type: Superiority; Hazard Ratio (HR) = 1.22, 95% CI 2-sided [0.85 to 1.73] — Stratified Cox proportional hazard model. Hazard Ratio is Nivolumab + Ipilimumab over Nivolumab

5. Secondary Outcome: Recurrence-free Survival (RFS) by Baseline Tumor PD-L1 Expression
Description: as for outcome 2
Time Frame: From randomization to Study Completion Date (up to approximately 45 months)
Population: All randomized participants with variable PD-L1 expression levels (see data table for details). PD-L1 expression levels based on clinical database.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Nivo + Ipi | Arm B: Nivo
Number analyzed (Participants) | 920 | 924
Months
  < 1% Tumor PD-L1 Expression: number analyzed (Participants) | 350 | 350
  < 1% Tumor PD-L1 Expression | 33.18 [22.21 to NA] — Upper limit not calculable as upper CI bound does not cross 50% threshold | 25.33 [19.81 to NA] — Upper limit not calculable as upper CI bound does not cross 50% threshold
  ≥ 1% Tumor PD-L1 Expression: number analyzed (Participants) | 527 | 534
  ≥ 1% Tumor PD-L1 Expression | NA [NA to NA] — Median not reached as Kaplan-Meier plot did not reach 0.5 probability of recurrence-free survival | NA [NA to NA] — Median not reached as Kaplan-Meier plot did not reach 0.5 probability of recurrence-free survival
  ≥ 5% Tumor PD-L1 Expression: number analyzed (Participants) | 300 | 303
  ≥ 5% Tumor PD-L1 Expression | NA [NA to NA] — Median not reached as Kaplan-Meier plot did not reach 0.5 probability of recurrence-free survival | NA [NA to NA] — Median not reached as Kaplan-Meier plot did not reach 0.5 probability of recurrence-free survival
  < 5% Tumor PD-L1 Expression: number analyzed (Participants) | 577 | 581
  < 5% Tumor PD-L1 Expression | NA [31.18 to NA] — Median not reached as Kaplan-Meier plot did not reach 0.5 probability of recurrence-free survival | NA [27.63 to NA] — Median not reached as Kaplan-Meier plot did not reach 0.5 probability of recurrence-free survival
  Non-quantifiable Tumor PD-L1 Expression: number analyzed (Participants) | 43 | 40
  Non-quantifiable Tumor PD-L1 Expression | NA [22.41 to NA] — Median not reached as Kaplan-Meier plot did not reach 0.5 probability of recurrence-free survival | NA [10.87 to NA] — Median not reached as Kaplan-Meier plot did not reach 0.5 probability of recurrence-free survival
Statistical Analysis 1: Comparison: Arm A: Nivo + Ipi vs Arm B: Nivo; Test type: Superiority — < 1% Tumor PD-L1 Expression; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.73 to 1.14] — Unstratisfied HR, Nivolumab over Ipilimumab
Statistical Analysis 2: Comparison: Arm A: Nivo + Ipi vs Arm B: Nivo; Test type: Superiority — >= 1% Tumor PD-L1 Expression; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.76 to 1.18] — Unstratisfied HR, Nivolumab over ipilimumab
Statistical Analysis 3: Comparison: Arm A: Nivo + Ipi vs Arm B: Nivo; Test type: Superiority — >= 5% Tumor PD-L1 Expression; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.71 to 1.34] — Unstratisfied HR, Nivolumab over ipilimumab
Statistical Analysis 4: Comparison: Arm A: Nivo + Ipi vs Arm B: Nivo; Test type: Superiority — < 5% Tumor PD-L1 Expression; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.77 to 1.10] — Unstratisfied HR, Nivolumab over ipilimumab
Statistical Analysis 5: Comparison: Arm A: Nivo + Ipi vs Arm B: Nivo; Test type: Superiority — Non-quantifiable Tumor PD-L1 Expression; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.38 to 1.51] — Unstratisfied HR, Nivolumab over ipilimumab

6. Secondary Outcome: Time to Next-Line Therapies - All Randomized Participants
Description: Time to next therapy was defined as the time from the date of randomization to the start date of next systemic therapy. Participants who did not receive next treatment were censored at the last known alive date.
  Time to second next therapy was defined as the time from the date of randomization to the start date of second next systemic therapy. Participants who did not receive second next treatment were censored at the last known alive date.
Time Frame: From randomization to start of next therapy or second next therapy (up to approximately 45 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Nivo + Ipi | Arm B: Nivo
Number analyzed (Participants) | 920 | 924
Months
  Time to next therapy | NA [NA to NA] — Median not reached because of an insufficient number of participants receiving next therapy | NA [NA to NA] — Median not reached because of an insufficient number of participants receiving next therapy
  Time to second next therapy | NA [NA to NA] — Median not reached because of an insufficient number of participants receiving second next therapy | NA [NA to NA] — Median not reached because of an insufficient number of participants receiving second next therapy

7. Secondary Outcome: Time to Next-Line Therapies - All Randomized Participants With PD-L1 Expression Level < 1%
Description: as for outcome 6
Time Frame: From randomization to start of next therapy or second next therapy (up to approximately 45 months)
Population: All randomized participants with PD-L1 expression level < 1%
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Nivo + Ipi | Arm B: Nivo
Number analyzed (Participants) | 349 | 351
Months
  Time to next therapy | NA [NA to NA] — Median not reached because of an insufficient number of participants receiving next therapy | NA [NA to NA] — Median not reached because of an insufficient number of participants receiving next therapy
  Time to second next therapy | NA [NA to NA] — Median not reached because of an insufficient number of participants receiving second next therapy | NA [NA to NA] — Median not reached because of an insufficient number of participants receiving second next therapy

8. Secondary Outcome: Time From Next Therapy to Second Next Therapy - All Randomized Participants
Description: Time from next treatment to second next treatment was defined as the time from the start date of next systemic therapy to start date of second next systemic therapy. No censoring rules were applied here as analysis was only performed for the subset of participants who received second next treatment.
Time Frame: From start of first next systemic therapy to start of second next systemic therapy (up to approximately 28 months)
Population: All randomized participants who received first and second next systemic therapy
Measure: Median (Full Range); unit: Months
Arm/Group | Arm A: Nivo + Ipi | Arm B: Nivo
Number analyzed (Participants) | 81 | 81
Months | 4.60 [0.8 to 23.7] | 4.80 [0.0 to 27.7]

9. Secondary Outcome: Time From Next Therapy to Second Next Therapy - All Randomized Participants With PD-L1 Expression Level < 1%
Description: as for outcome 8
Time Frame: From start of first next systemic therapy to start of second next systemic therapy (up to approximately 28 months)
Population: All randomized participants with PD-L1 expression level < 1% who received first and second next therapy
Measure: Median (Full Range); unit: Months
Arm/Group | Arm A: Nivo + Ipi | Arm B: Nivo
Number analyzed (Participants) | 35 | 46
Months | 4.44 [0.8 to 23.7] | 5.04 [0.9 to 27.7]

10. Secondary Outcome: Progression-free Survival (PFS) on Next-line Therapy - All Randomized Participants
Description: PFS2 was defined as the time from randomization to the progression date on next-line systemic therapy or the end date of next-line systemic therapy (if progression date not available) or death from any cause (if both progression date and end date not available), and to last known alive date in case of no event (ie, censoring), meaning either (1) no subsequent systemic therapy and no death OR (2) subsequent systemic therapy but no progression date nor end date available and no death.
Time Frame: From randomization to progression event (up to approximately 45 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Nivo + Ipi | Arm B: Nivo
Number analyzed (Participants) | 920 | 924
Months | NA [NA to NA] — Median not reached as insufficient progression events among participants | NA [NA to NA] — Median not reached as insufficient progression events among participants

11. Secondary Outcome: Progression-free Survival (PFS) on Next-line Therapy - All Randomized Participants With PD-L1 Expression Level < 1%
Description: as for outcome 10
Time Frame: From randomization to progression event (up to approximately 45 months)
Population: All randomized participants with PD-L1 expression level < 1%.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Nivo + Ipi | Arm B: Nivo
Number analyzed (Participants) | 349 | 351
Months | NA [NA to NA] — Median not reached as insufficient progression events among participants | NA [35.94 to NA] — Median not reached as insufficient progression events among participants

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from first dose to study completion date (up to approximately 45 months). Serious Adverse Events and Non Serious Adverse Events above 5% were assessed from first dose to 100 days post last dose (up to approximately 15 months)
Arm/Group | Arm A: Nivo + Ipi | Arm B: Nivo
All-Cause Mortality (participants affected / at risk) | 122/916 | 121/917
Serious Adverse Events (participants affected / at risk) | 374/916 | 242/917
Other Adverse Events (participants affected / at risk) | 868/916 | 844/917
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Nivo + Ipi (N=916) | Arm B: Nivo (N=917)
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 3
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Splenic lesion (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 4 | 0
Atrial flutter (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardio-respiratory distress (Cardiac disorders) | 1 | 0
Cardiomegaly (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Myocarditis (Cardiac disorders) | 3 | 0
Palpitations (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Addison's disease (Endocrine disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 10 | 2
Adrenocortical insufficiency acute (Endocrine disorders) | 0 | 1
Adrenocorticotropic hormone deficiency (Endocrine disorders) | 0 | 1
Goitre (Endocrine disorders) | 0 | 1
Hyperparathyroidism (Endocrine disorders) | 0 | 1
Hyperparathyroidism primary (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 5 | 0
Hypophysitis (Endocrine disorders) | 24 | 9
Hypothyroidism (Endocrine disorders) | 2 | 1
Lymphocytic hypophysitis (Endocrine disorders) | 3 | 0
Primary adrenal insufficiency (Endocrine disorders) | 1 | 0
Thyroiditis (Endocrine disorders) | 2 | 1
Thyroiditis acute (Endocrine disorders) | 1 | 1
Thyrotoxic crisis (Endocrine disorders) | 1 | 0
Orbital myositis (Eye disorders) | 1 | 1
Papilloedema (Eye disorders) | 0 | 2
Retinal detachment (Eye disorders) | 0 | 1
Retinal tear (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Autoimmune colitis (Gastrointestinal disorders) | 8 | 2
Autoimmune pancreatitis (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 29 | 7
Colitis microscopic (Gastrointestinal disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 18 | 7
Duodenitis (Gastrointestinal disorders) | 1 | 1
Enteritis (Gastrointestinal disorders) | 1 | 1
Enterocolitis (Gastrointestinal disorders) | 2 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 2 | 0
Gastritis (Gastrointestinal disorders) | 4 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Immune-mediated enterocolitis (Gastrointestinal disorders) | 16 | 7
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Oesophageal obstruction (Gastrointestinal disorders) | 1 | 0
Oesophageal spasm (Gastrointestinal disorders) | 1 | 0
Pancreatic cyst (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 4
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 | 1
Retroperitoneal fibrosis (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0
Ulcerative gastritis (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Complication associated with device (General disorders) | 0 | 1
Fatigue (General disorders) | 6 | 0
Gait disturbance (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 1 | 0
Granuloma (General disorders) | 1 | 0
Lithiasis (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Mass (General disorders) | 1 | 0
Nodule (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Polyserositis (General disorders) | 0 | 1
Pyrexia (General disorders) | 12 | 5
Autoimmune hepatitis (Hepatobiliary disorders) | 14 | 1
Cholangitis sclerosing (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 6 | 4
Hepatotoxicity (Hepatobiliary disorders) | 4 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1
Immune-mediated hepatitis (Hepatobiliary disorders) | 6 | 0
Liver disorder (Hepatobiliary disorders) | 2 | 1
Nodular regenerative hyperplasia (Hepatobiliary disorders) | 1 | 0
Venoocclusive liver disease (Hepatobiliary disorders) | 1 | 0
Autoimmune disorder (Immune system disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Sarcoidosis (Immune system disorders) | 7 | 1
Adrenalitis (Infections and infestations) | 1 | 2
Arthritis bacterial (Infections and infestations) | 0 | 1
Atypical pneumonia (Infections and infestations) | 3 | 0
Bacterial infection (Infections and infestations) | 1 | 0
Bronchiolitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 2
Bronchitis viral (Infections and infestations) | 1 | 0
Bursitis infective (Infections and infestations) | 2 | 0
Campylobacter colitis (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 4 | 5
Chronic sinusitis (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Cytomegalovirus infection reactivation (Infections and infestations) | 0 | 1
Dengue fever (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 1 | 0
Diarrhoea infectious (Infections and infestations) | 1 | 0
Encephalitis (Infections and infestations) | 4 | 2
Endocarditis enterococcal (Infections and infestations) | 1 | 0
Enterovirus infection (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 5 | 3
Fournier's gangrene (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 1
Groin abscess (Infections and infestations) | 1 | 0
Haematoma infection (Infections and infestations) | 0 | 1
Herpes oesophagitis (Infections and infestations) | 1 | 0
Infected bite (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 3 | 1
Meningitis (Infections and infestations) | 2 | 0
Meningitis aseptic (Infections and infestations) | 2 | 0
Myelitis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Picornavirus infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 11 | 2
Pneumonia klebsiella (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 3 | 0
Septic shock (Infections and infestations) | 2 | 1
Sinusitis (Infections and infestations) | 1 | 1
Skin infection (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 2
Tonsillitis (Infections and infestations) | 1 | 0
Tracheitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 1
Urosepsis (Infections and infestations) | 3 | 0
Varicella zoster virus infection (Infections and infestations) | 0 | 1
Vascular device infection (Infections and infestations) | 1 | 1
Vestibular neuronitis (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Graft complication (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 3
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic liver injury (Injury, poisoning and procedural complications) | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 2
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 0
Amylase increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Electrocardiogram abnormal (Investigations) | 1 | 0
General physical condition abnormal (Investigations) | 1 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Lipase increased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 2 | 1
Troponin I increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 1
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 | 0
Fulminant type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2
Steroid diabetes (Metabolism and nutrition disorders) | 4 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 2
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 2 | 2
Myositis-like syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 2 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 | 23
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 7
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 | 10
Marginal zone lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Melanoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 1
Metastases to breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Recurrent cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 12
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute disseminated encephalomyelitis (Nervous system disorders) | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0
Autoimmune neuropathy (Nervous system disorders) | 1 | 0
Carotid artery dissection (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Encephalitis autoimmune (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 2 | 0
Epilepsy (Nervous system disorders) | 0 | 1
Facial paresis (Nervous system disorders) | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 4
Hypertensive encephalopathy (Nervous system disorders) | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 1 | 0
Meningism (Nervous system disorders) | 0 | 1
Miller Fisher syndrome (Nervous system disorders) | 1 | 0
Monoparesis (Nervous system disorders) | 1 | 0
Myasthenia gravis (Nervous system disorders) | 2 | 0
Myasthenic syndrome (Nervous system disorders) | 0 | 1
Myelitis transverse (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Optic neuritis (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0
Radiculopathy (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 2 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 2 | 3
Mania (Psychiatric disorders) | 1 | 0
Mental disorder (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 4 | 4
Autoimmune nephritis (Renal and urinary disorders) | 0 | 2
Calculus bladder (Renal and urinary disorders) | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Nephritis (Renal and urinary disorders) | 1 | 3
Nephrolithiasis (Renal and urinary disorders) | 2 | 0
Renal colic (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 2 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diaphragmatic spasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Immune-mediated pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 9 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 1
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 | 2
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 2 | 1
Capillary leak syndrome (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 1
Hypertension (Vascular disorders) | 2 | 1
Lymphoedema (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
Shock (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Nivo + Ipi (N=916) | Arm B: Nivo (N=917)
Adrenal insufficiency (Endocrine disorders) | 56 | 7
Hyperthyroidism (Endocrine disorders) | 180 | 98
Hypophysitis (Endocrine disorders) | 92 | 11
Hypothyroidism (Endocrine disorders) | 219 | 139
Abdominal pain (Gastrointestinal disorders) | 102 | 84
Abdominal pain upper (Gastrointestinal disorders) | 57 | 37
Constipation (Gastrointestinal disorders) | 108 | 89
Diarrhoea (Gastrointestinal disorders) | 338 | 304
Dry mouth (Gastrointestinal disorders) | 99 | 90
Nausea (Gastrointestinal disorders) | 218 | 187
Vomiting (Gastrointestinal disorders) | 100 | 77
Asthenia (General disorders) | 165 | 147
Fatigue (General disorders) | 348 | 338
Influenza like illness (General disorders) | 58 | 47
Pyrexia (General disorders) | 118 | 84
Nasopharyngitis (Infections and infestations) | 109 | 101
Upper respiratory tract infection (Infections and infestations) | 69 | 86
Infusion related reaction (Injury, poisoning and procedural complications) | 56 | 46
Alanine aminotransferase increased (Investigations) | 134 | 86
Amylase increased (Investigations) | 85 | 37
Aspartate aminotransferase increased (Investigations) | 110 | 70
Blood creatine phosphokinase increased (Investigations) | 56 | 50
Lipase increased (Investigations) | 120 | 58
Decreased appetite (Metabolism and nutrition disorders) | 106 | 63
Hyperglycaemia (Metabolism and nutrition disorders) | 51 | 49
Arthralgia (Musculoskeletal and connective tissue disorders) | 168 | 213
Back pain (Musculoskeletal and connective tissue disorders) | 94 | 96
Myalgia (Musculoskeletal and connective tissue disorders) | 99 | 81
Pain in extremity (Musculoskeletal and connective tissue disorders) | 47 | 52
Dizziness (Nervous system disorders) | 67 | 64
Headache (Nervous system disorders) | 270 | 214
Anxiety (Psychiatric disorders) | 32 | 47
Insomnia (Psychiatric disorders) | 88 | 75
Cough (Respiratory, thoracic and mediastinal disorders) | 162 | 168
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 73 | 74
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 52 | 43
Pruritus (Skin and subcutaneous tissue disorders) | 339 | 238
Rash (Skin and subcutaneous tissue disorders) | 258 | 234
Vitiligo (Skin and subcutaneous tissue disorders) | 49 | 56
Hypertension (Vascular disorders) | 42 | 47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-03-11): https://cdn.clinicaltrials.gov/large-docs/55/NCT03068455/Prot_002.pdf
  • Statistical Analysis Plan (2019-08-23): https://cdn.clinicaltrials.gov/large-docs/55/NCT03068455/SAP_003.pdf